CLINICAL TRIAL: NCT04137003
Title: Laval University Rouge et Or Post Anterior Cruciate Ligament Surgery Readaptation Program Effectiveness With Amateur Athletes: A Randomised Clinical Trial
Brief Title: Laval University Rouge et or Post ACL Surgery Program Effectiveness
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Laval University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ACL readaptation LavalU
Record Dates: First submitted 2019-07-03; First posted 2019-10-23 (Actual); Last update posted 2019-10-28 (Actual); Status verified 2019-10

CONDITIONS: Anterior Cruciate Ligament Injuries; ACL
Keywords: Acl; Anterior cruciate ligament; Post surgery
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Intervention Model Description: Experimental research with pre-post repeated measures with a control group. It is a randomised control trial with a blinded assessor
Who Masked: Outcomes Assessor
Masking Description: Subjects are randomised to one of the two groups: Rouge et or program or Chu protocol. The assessor that perform the multiple assessments is blinded to the randomisation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rouge et Or program (Experimental): Rouge et Or program group follow a detailed program that they do on their own. It is made of three cycles of four weeks each. Every cycle contains 3 training sessions by week with a minimum of 24 hours between sessions. The training volume is modulated for every cycle and every week. Each training sessions is made of 6 warm-up exercises followed by 6 training exercises. The exercises are a mix of strengthening, endurance, plyometric, neuromuscular control and dynamic stability. The exercises change every month with a progressively increasing difficulty towards the end to mimic return to sport demands.
  Interventions: Other: Rouge et Or Program
- CHU intervention guide (Active Comparator): CHU intervention guide group follow the standard CHU protocol. At three months post-surgery, the protocol suggests progressing the exercises without precisely suggesting exercise, parameter or frequency.
  Interventions: Other: CHU intervention guide

INTERVENTIONS:
Other: Rouge et Or Program — It is a detailed, structured and precise training program. It is used from the third-month post ACL surgery to the sixth month.
  Other Names: (Gr PRORO-UL); Programme du rouge et Or; Laval University Rouge et Or program
  Arms: Rouge et Or program
Other: CHU intervention guide — From the third month to the sixth month, it outlines the progression to have in the training without precise information on exercises, parameter or frequency.
  Other Names: Programme du CHU; (Gr CHU-CP); CHU program
  Arms: CHU intervention guide

SUMMARY:
The main objective is to compare the effectiveness of two readaptation programs post anterior cruciate ligament surgery. Laval University Rouge et or program is to be compared with the intervention guide from the CHU. Amateur athletes are recruited 3 months post ACL surgery. The level of confidence, symptoms, functional recovery level and muscle strength are assessed and compared between the two groups at 3, 4, 5, 6 and 9-month post surgery.

DETAILED DESCRIPTION:
It is experimental research with pre-post repeated measure with a control group. The subjects are randomised either in the intervention group (Gr PRORO-UL) or the control group (Gr CHU-CP). The assessor is blinded to the randomisation. Both groups receive their program at the first assessment at three months post-ACL-surgery. They are strongly encouraged to continue their follow-up in physiotherapy to ensure the program is suitable to their individual progression. The participants are assessed again at 4, 5, 6 and 9 months post surgery to measure their progression. A weekly journal sent by e-mail is to be filled to ensure the subjects train according to their program attribution. It is a randomised control trial with a blinded assessor.

ELIGIBILITY:
Inclusion Criteria:

* Amateur athlete aged from 18 to 35 years old doing sports at least 3 times a week
* Having suffered from an Anterior Cruciate Ligament rupture
* Having undergone Anterior Cruciate Ligament surgery either with an anterior approach (with the patellar tendon) or a posterior approach (with the semitendinosus tendon)
* Having a functional deficit (score 85% or under at Knee Outcome Survey - Activity of Daily Living Scale questionnaire and/or score 80% or under at International Knee Documentation Committee questionnaire)
* Being available for follow up and actively follow the programme attributed.

Exclusion Criteria:

* Having suffered from multiple surgery for other ligaments in the same knee.
* Having undergone total meniscus removal
* Having suffered form Posterior Cruciate Ligament rupture.
* Having other injuries that could affect the functional performance and prevent from training.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-03-06 (Actual); Primary Completion 2020-09-01 (Estimated); Study Completion 2020-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in Knee Outcome Survey-Activity of Daily Living Scale | 3, 4, 5, 6 and 9 months post-surgery
  Questionnaire ranging from 0 to 70 over 70 where 70 means no limitation in activity of daily living. There is 14 questions with each graded answer providing 0 to 5 points that are summed together and expressed in percentage. The higher is the score, the better is the outcome.

SECONDARY OUTCOMES:
Numerical Pain Rating Scale | 3 months post surgery
  Four questions related to pain that are graded from 0 to 10. The lower is the score, the better is the outcome.
Numerical Pain Rating Scale | 4 months post-surgery
  Four questions related to pain that are graded from 0 to 10. The lower is the score, the better is the outcome.
Numerical Pain Rating Scale | 5 months post-surgery
  Four questions related to pain that are graded from 0 to 10. The lower is the score, the better is the outcome.
Numerical Pain Rating Scale | 6 months post-surgery
  Four questions related to pain that are graded from 0 to 10. The lower is the score, the better is the outcome.
Numerical Pain Rating Scale | 9 months post-surgery
  Four questions related to pain that are graded from 0 to 10. The lower is the score, the better is the outcome.
Change in Anterior Cruciate Ligament Return to Sport Index | 3, 4, 5, 6 and 9 months post-surgery
  12 questions related to return to sport confidence graded from 0 to 10. All scores are summed together and expressed in percentage.The higher the score the better is the outcome.
Change in International knee documentation committee | 3, 4, 5, 6 and 9 months post-surgery
  International knee documentation committee is a 10 items questionnaire measuring knee functional limitation. All items are summed and the total score range from 18 to 105. From that score we subtract 18 and divide by 87 and bring the score back in percentage. The final score can range from 0 to 100% where a higher score represents a better outcome.
Muscle strength | 3 months post-surgery
  Isometric flexion and extension strength is measured with a handheld dynamometer.
Muscle strength | 4 months post-surgery
  Isometric flexion and extension strength is measured with a handheld dynamometer.
Muscle strength | 5 months post-surgery
  Isometric flexion and extension strength is measured with a handheld dynamometer.
Muscle strength | 6 months post-surgery
  Isometric flexion and extension strength is measured with a handheld dynamometer.
Muscle strength | 9 months post-surgery
  Isometric flexion and extension strength is measured with a handheld dynamometer.
Muscle strength | 6 months post-surgery.
  Concentric isokinetic flexion and extension strength is measured with Biodex at speed 60 degree/sec.
Muscle strength | 9 months post-surgery.
  Concentric isokinetic flexion and extension strength is measured with Biodex at speed 60 degree/sec.
Single leg hop test. | 3 months post-surgery
  The single-leg hop test is performed barefoot. The subjects are asked to jump as far as possible on one leg and to land keeping their balance. Measurement is made from the starting line to the place where the heel lands. The subjects must start behind the line. They perform one practice and three trials. The best trial is kept. The healthy limb is tested first followed by the injured leg.
Single leg hop test. | 4 months post-surgery
  The single-leg hop test is performed barefoot. The subjects are asked to jump as far as possible on one leg and to land keeping their balance. Measurement is made from the starting line to the place where the heel lands. The subjects must start behind the line. They perform one practice and three trials. The best trial is kept. The healthy limb is tested first followed by the injured leg.
Single leg hop test. | 5 months post-surgery
  The single-leg hop test is performed barefoot. The subjects are asked to jump as far as possible on one leg and to land keeping their balance. Measurement is made from the starting line to the place where the heel lands. The subjects must start behind the line. They perform one practice and three trials. The best trial is kept. The healthy limb is tested first followed by the injured leg.
Single leg hop test. | 6 months post-surgery
  The single-leg hop test is performed barefoot. The subjects are asked to jump as far as possible on one leg and to land keeping their balance. Measurement is made from the starting line to the place where the heel lands. The subjects must start behind the line. They perform one practice and three trials. The best trial is kept. The healthy limb is tested first followed by the injured leg.
Single leg hop test. | 9 months post-surgery
  The single-leg hop test is performed barefoot. The subjects are asked to jump as far as possible on one leg and to land keeping their balance. Measurement is made from the starting line to the place where the heel lands. The subjects must start behind the line. They perform one practice and three trials. The best trial is kept. The healthy limb is tested first followed by the injured leg.
Triple hop test. | 3 months post-surgery
  The Triple hop test is performed barefoot. The subjects are asked to jump on one leg three times in a row in one direction and to land the third jump in balance as far as possible. Measurement is made from the starting line to the place where the heel lands the third jump. The subjects must start behind the line. They perform one practice and three trial. The best trial is kept. The healthy limb is tested first followed by the injured leg.
Triple hop test. | 4 months post-surgery
  The Triple hop test is performed barefoot. The subjects are asked to jump on one leg three times in a row in one direction and to land the third jump in balance as far as possible. Measurement is made from the starting line to the place where the heel lands the third jump. The subjects must start behind the line. They perform one practice and three trial. The best trial is kept. The healthy limb is tested first followed by the injured leg.
Triple hop test. | 5 months post-surgery
  The Triple hop test is performed barefoot. The subjects are asked to jump on one leg three times in a row in one direction and to land the third jump in balance as far as possible. Measurement is made from the starting line to the place where the heel lands the third jump. The subjects must start behind the line. They perform one practice and three trial. The best trial is kept. The healthy limb is tested first followed by the injured leg.
Triple hop test. | 6 months post-surgery
  The Triple hop test is performed barefoot. The subjects are asked to jump on one leg three times in a row in one direction and to land the third jump in balance as far as possible. Measurement is made from the starting line to the place where the heel lands the third jump. The subjects must start behind the line. They perform one practice and three trial. The best trial is kept. The healthy limb is tested first followed by the injured leg.
Triple hop test. | 9 months post-surgery
  The Triple hop test is performed barefoot. The subjects are asked to jump on one leg three times in a row in one direction and to land the third jump in balance as far as possible. Measurement is made from the starting line to the place where the heel lands the third jump. The subjects must start behind the line. They perform one practice and three trial. The best trial is kept. The healthy limb is tested first followed by the injured leg.
30 seconds side hop test | 3 months post-surgery
  The 30 seconds side hop test is performed barefoot. The subjects are asked to jump side to side on one leg as many time as possible during 30 seconds over a 40 cm distance separated by two lines. Each time the foot of the subjet touch one line, the repetition is not recorded. The number of jumps is recorded. They perform two practice jumps and one 30 secondes trial. The healthy limb is tested first followed by the injured leg.
30 seconds side hop test | 4 months post-surgery
  The 30 seconds side hop test is performed barefoot. The subjects are asked to jump side to side on one leg as many time as possible during 30 seconds over a 40 cm distance separated by two lines. Each time the foot of the subjet touch one line, the repetition is not recorded. The number of jumps is recorded. They perform two practice jumps and one 30 secondes trial. The healthy limb is tested first followed by the injured leg.
30 seconds side hop test | 5 months post-surgery
  The 30 seconds side hop test is performed barefoot. The subjects are asked to jump side to side on one leg as many time as possible during 30 seconds over a 40 cm distance separated by two lines. Each time the foot of the subjet touch one line, the repetition is not recorded. The number of jumps is recorded. They perform two practice jumps and one 30 secondes trial. The healthy limb is tested first followed by the injured leg.
30 seconds side hop test | 6 months post-surgery
  The 30 seconds side hop test is performed barefoot. The subjects are asked to jump side to side on one leg as many time as possible during 30 seconds over a 40 cm distance separated by two lines. Each time the foot of the subjet touch one line, the repetition is not recorded. The number of jumps is recorded. They perform two practice jumps and one 30 secondes trial. The healthy limb is tested first followed by the injured leg.
30 seconds side hop test | 9 months post-surgery
  The 30 seconds side hop test is performed barefoot. The subjects are asked to jump side to side on one leg as many time as possible during 30 seconds over a 40 cm distance separated by two lines. Each time the foot of the subjet touch one line, the repetition is not recorded. The number of jumps is recorded. They perform two practice jumps and one 30 secondes trial. The healthy limb is tested first followed by the injured leg.
Global Rating Of Change | 4 months post-surgery
  A 15 item scale to grade the change from the initial data collection.
Global Rating Of Change | 5 post-surgery
  A 15 item scale to grade the change from the initial data collection.
Global Rating Of Change | 6 post-surgery
  A 15 item scale to grade the change from the initial data collection.
Global Rating Of Change | 9 post-surgery
  A 15 item scale to grade the change from the initial data collection.

CONTACTS AND LOCATIONS:
Overall Officials: Luc J. Hébert, PHD, Study Director — Laval University
Locations (1):
- Université Laval, Québec, Canada

IPD SHARING:
Plan to Share IPD: No